CLINICAL TRIAL: NCT04478344
Title: Precise Ultrasound Localization and Guided Injection for Superior Cluneal Nerve Entrapment
Brief Title: Ultrasound Localization and Guided Injection for Superior Cluneal Nerve Entrapment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201912037RINC
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain; Nerve Entrapment Syndrome
Keywords: Ultrasonography; Superior cluneal nerve; Nerve entrapment; Prediction; Ultrasound-guided injection; Hydrodissection
MeSH Terms: conditions — Low Back Pain; Charcot-Marie-Tooth Disease; Nerve Compression Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided hydrodissection to superior cluneal nerve (Experimental): Patients with superior cluneal nerve enttrappment given by ultrasound guided perineural injection with a mixture of 1 mL of 50% dextrose, 4 mL of 1% lidocaine, and 5 mL of 0.9% normal saline to superior cluneal nerve of affected side.
  Interventions: Other: Ultrasound guided hydrodissection of superior cluneal nerve
- Control arm (No Intervention): Patients without superior cluneal nerve entrappment

INTERVENTIONS:
Other: Ultrasound guided hydrodissection of superior cluneal nerve — Intervention procedure: hydrodissection to the superior cluneal nerve entrapment; Device for guidance of injection: high-resolution ultrasound ; Drug for injection: a mixture of 1 mL of 50% dextrose, 4 mL of 1% lidocaine, and 5 mL of 0.9% normal saline
  Arms: Ultrasound guided hydrodissection to superior cluneal nerve

SUMMARY:
Low back pain (LBP) is a common complaint in the clinical setting. Among all the differential diagnosis for LBP, superior cluneal nerve (SCN) entrapment is the commonly omitted one. The superior cluneal nerve is the terminal branch of the lateral branches of the posterior rami of the L1-L3 spinal nerves, which passes through the osseous tunnel interposed between the thoracolumbar fascia and iliac crest. This nerve can be entrapped due to poor posture, trauma or stretching of the surrounding thoracolumbar fascia and osseous membrane. The cardinal symptom of the superior cluneal nerve entrapment is buttock pain. Sometimes the pain may radiate to the lower limb, which mimics sciatica, and makes the diagnosis difficult. Early diagnosis and treatment of SCN entrapment is crucial, which can facilitate the improvement of health related quality of life and decrement the socioeconomic loss due to disability.

The study aims is (1) to scan the SCN and thoracolumbar fascia by ultrasound in patients with LBP and normal subjects. The transcutaneous electrical stimulation will be used to confirm the location of SCN by asking the subject to depict the sensory distribution after stimulation; (2) to analyze the related factors of LBP with SCN entrapment, which may help in setting up the diagnostic criteria of SCN entrapment; (3) to analyze the therapeutic effect of perineural injection to SCN in SCN entrapment, and to find the factors that related responsiveness.

DETAILED DESCRIPTION:
Introduction:

Superior cluneal nerve (SCN) entrapment is the commonly omitted diagnosis in chronic low back pain. The superior cluneal nerve is the terminal branch of the lateral branches of the posterior rami of the L1-L3 spinal nerves, which passes through the osseous tunnel interposed between the thoracolumbar fascia and iliac crest. This nerve can be entrapped due to poor posture, trauma or stretching of the surrounding thoracolumbar fascia and osseous membrane. The cardinal symptom of the superior cluneal nerve entrapment is buttock pain. Sometimes the pain may radiate to the lower limb, which mimics sciatica, and makes the diagnosis difficult. Early diagnosis and treatment of SCN entrapment is crucial, which can facilitate the improvement of health related quality of life and decrement the socioeconomic loss due to disability.

Material and methods:

Participants: Adult patients (>20 year old) with low back/buttock pain. The pain consists area of iliac crest.

Control : healthy adult subjects (>20 year old) without low back

Exclusion criteria: non-mechanical low back pain, referred low back pain (tumor, infection, inflammatory arthritis, Scheuermann disease,Paget disease, herpetic neuralgia), trauma, acute compression fracture, acute herniated disc, underwent nerve block within 3 months.

Study design:

(1) To scan the SCN and thoracolumbar fascia by high-resolution ultrasound in patients with LBP and normal subjects. The transcutaneous electrical stimulation will be used to confirm the location of SCN by asking the subject to depict the sensory distribution after stimulation; (2) to analyze the related factors of LBP with SCN entrapment, which may help in setting up the diagnostic criteria of SCN entrapment; (3) to analyze the therapeutic effect of perineural injection to SCN in SCN entrapment, and to find the factors that related responsiveness.

Detail of the intervention

1. High-resolution ultrasound evaluation of buttock region to recognize the superior cluneal nerve in patients with SCN entrapment and healthy control. The transcutaneous electrical stimulation will be assisted device for confirming the diagnosis by subjective response of patients.
2. Collecting the LBP-related information, including physical examination results ((SLRT, Extension in one-leg standing, Gaeslen's test, Yeoman's test, compression test, distraction test, FABER test and ROM), lumbosacral and pelvic X-ray. Compare the related information with sonography results.
3. Intervention: single arm experiment design. Ultrasound guided perineural injection with 1 mL of 50% dextrose, 4 mL of 1% lidocaine, and 5 mL of 0.9 % normal saline to the site where SCN being entrapment, to evaluate the clinical efficacy of perineural injection to SCN entrapment.

Outcome measurement:

Primary outcome :

1. Visual analogue scale
2. Modified version of the Oswestry Disability Questionnaire used in the AAOS lumbar cluster
3. Short-Form-36 (SF-36)

at baseline one month and three months after injection

Secondary outcome:

1. Sonography (gray-scale/elastography) at baseline, one month and three months after injection
2. Pressure pain threshold

Statistical analysis:

Continuous variables

1. Student's t test: fit assumption of normal distribution
2. Mann-Whitney test: does not fit the assumption of normal distribution Categorical variables

1. Chi-square test 2. Fisher exact test: sparse data

Multivariate analysis:

Generalized Estimating Equations

ELIGIBILITY:
Participants:

* Adult patients (>20 year old) with low back/buttock pain.
* The pain consists area of iliac crest Control : healthy adult subjects (>20 year old) without low back

Exclusion criteria:

* non-mechanical low back pain
* referred low back pain (tumor, infection, inflammatory arthritis, Scheuermann disease,Paget disease, herpetic neuralgia)
* trauma
* acute compression fracture
* acute herniated disc
* underwent lumbar region nerve block within 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Questionnaire | Change of the score between one month and baseline, and change of the score between three months and baseline
  Oswestry Disability Questionnaire, A 10 item questionnaire, score ranges from 0 to 100, and a higher score indicates worse function.
Short Form-36 Questionnaire | Change of the score between one month and baseline, and change of the score between three month and baseline
  Reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social func-tion, emotional role, and mental health. The categories of physical role and emotional role reflect performance at the activity and participation levels. The score will be transformed between 0 to 100. The higher score means better health condition in each domain.
Visual analogue scale | Change of the score between one month and baseline, and change of the score between three months and baseline
  The pain scale to evaluate pain, from 0 to 10. The lower means less pain.

SECONDARY OUTCOMES:
Ultrasound evaluation of SCN (Grey scale) | Measurement change between one month and baseline and between three months and baseline
  Measurement of cross sectional area (square millimeters) and record image

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Vin Chang, MD,PhD, Principal Investigator — National Taiwan University Hospital Bei-Hu Branch
Locations (1):
- National Taiwan University Hospital, Bei-Hu Branch, Taipei, Wanhua District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu WT, Mezian K, Nanka O, Chen LR, Ricci V, Lin CP, Chang KV, Ozcakar L. Enhancing diagnosis and treatment of superior cluneal nerve entrapment: cadaveric, clinical, and ultrasonographic insights. Insights Imaging. 2023 Jul 3;14(1):116. doi: 10.1186/s13244-023-01463-0. PMID 37395948